CLINICAL TRIAL: NCT06498765
Title: Effect of Pacifier Use During Phototherapy on Stress and Bilirubin Level in Newborns With Hyperbilirubinemia
Brief Title: Pacifier Use During Phototherapy in Newborns With Hyperbilirubinemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Ahu Pınar TURAN, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC
Record Dates: First submitted 2024-06-29; First posted 2024-07-12 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Newborn Jaundice; Pacifier
Keywords: newborn; pacifier; stress; bilirubinemia; phototherapy
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The newborns in the experimental group were given a pacifier.
  Interventions: Other: Pacifier Use
- Control group (No Intervention): The newborns in the control group were not given a pacifier.

INTERVENTIONS:
Other: Pacifier Use — The newborns in the experimental group were given a pacifier, unlike the control group. The newborns were placed in a phototherapy incubator and each time they were placed in a phototherapy incubator, the newborns were given a pacifier for an average of 5 minutes. The researcher encouraged the babies to take the pacifier.
  Arms: Experimental group

SUMMARY:
Hyperbilirubinemia; It is a common condition that usually occurs physiologically in newborns. Phototherapy is used in the treatment of hyperbilirubinemia. Babies cry while receiving phototherapy, the mother's inability to hold her baby in her arms, her inability to breastfeed, and the invasive procedures (bloodletting) stress the baby. Pacifiers are used among individualized developmental care practices to calm the baby and reduce stress. Another benefit of pacifiers for the baby is on the gastrointestinal system. Non-nutritive sucking stimulates oro-motor development, facilitates the development of sucking behavior and facilitates digestion in enteral feeding. Considering all these benefits, this study aimed to determine the effect of pacifier use during phototherapy on stress and bilirubin levels in newborns with hyperbilirubinemia.

DETAILED DESCRIPTION:
After birth, fetal erythrocytes in the newborn are rapidly destroyed and the total bilirubin level increases, resulting in hyperbilirubinemia. Hyperbilirubinemia; although it is a common condition that usually occurs physiologically in newborns, it causes neurological dysfunction in the newborn when it reaches high bilirubin levels. Therefore, follow-up and treatment are important. One of the treatment approaches for hyperbilirubinemia is phototherapy.

Phototherapy treatment is applied to babies diagnosed with hyperbilirubinemia by directly giving light energy to the babies. While receiving phototherapy, the baby becomes stressed due to reasons such as the mother not being able to hold her baby in her arms, not being able to breastfeed, the baby being in a different environment such as the neonatal intensive care unit, and being exposed to invasive procedures. Individualized developmental care practices accordingly, many practices are recommended in neonatal intensive care units to reduce the stress of babies. One of these practices is non-nutritive sucking. The most commonly used method for non-nutritive sucking is the use of a pacifier. It is stated that the use of pacifiers helps the baby calm down and reduces stress in neonatal intensive care units. In 1990, the World Health Organization and the United Nations International Children's Emergency Fund determined the "Ten Steps to Successful Breastfeeding" principles for the Baby-Friendly Hospital Initiative to promote and support breastfeeding. It has been noticed that in these principles rejecting the use of pacifiers, intensive care environments where the baby is stressed and situations where the mother and the baby are separated are ignored, so it has been suggested that this situation should be brought back to the agenda. In 2013, the "Ten Steps to Successful Breastfeeding" application was revised; Considering the justified reasons for the special situations in which the newborn and the mother and the baby are separated and the situations in which the baby is stressed, the newborn The use of pacifiers has been recommended in intensive care units. Considering the 24-hour treatment period during phototherapy, the baby is separated from the mother, albeit intermittently, while receiving phototherapy. In addition, the baby is in a different environment such as the neonatal intensive care unit and is exposed to invasive procedures. All of these create stress in the baby, and pacifiers are recommended for such justified reasons. The benefits of pacifier use have been proven in neonatal intensive care units, such as calming the baby, making it easier to fall asleep, and reducing pain and stress. Another benefit of non-nutritive sucking is on the gastrointestinal system. Non-nutritive sucking stimulates oro-motor development, facilitates the development of sucking behavior and facilitates digestion in enteral feeding.

A number of enzymes and hormones are involved in facilitating digestion through non-nutritive absorption. These enzymes and hormones; lingual lipase, gastrin, insulin and motilin. Experts believe that non-nutritive sucking causes this effect through vagal stimulation of the oral mucosa. It is thought that it causes the secretion of enzymes and hormones. Non-nutritive sucking in a study reported that the use of pacifiers, one of the methods, stimulates the stomach motor functions and this facilitates the digestive process through the activation of vagal mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns
* Newborns diagnosed with hyperbilirubinemia
* Babies who do not use pacifiers
* Newborns scheduled to receive phototherapy for 24 hours
* Babies of parents who agreed to participate in the study

Exclusion Criteria:

* Newborns receiving other treatments along with phototherapy
* Newborns with a diagnosis other than hyperbilirubinemia
* Newborns using antibiotics
* Babies fed with formula milk or bottle
* Babies diagnosed with pathological Hyperbilirubinemia

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate peak | mother's arms, 5 minutes after the baby is placed in the phototherapy bed, 5 minutes after the baby is placed in the phototherapy bed at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours.
  The heart rate of the baby receiving phototherapy was measured with a pulse oximeter device attached to the baby's wrist. The evaluation will be done while the baby is in the mother's arms, 5 minutes after being placed on the phototherapy bed, and at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st and 24th hours after being placed on the phototherapy bed.
Oxygen saturation | mother's arms, 5 minutes after the baby is placed in the phototherapy bed, 5 minutes after the baby is placed in the phototherapy bed at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours.
  The oxygen saturation of the baby receiving phototherapy was measured with a pulse oximeter device attached to the baby's wrist. The evaluation will be done while the baby is in the mother's arms, 5 minutes after being placed on the phototherapy bed, and at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st and 24th hours after being placed on the phototherapy bed.
Bowel sounds | mother's arms, 5 minutes after the baby is placed in the phototherapy bed, 5 minutes after the baby is placed in the phototherapy bed at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours.
  The bowel sounds of the baby receiving phototherapy was measured with a pulse oximeter device attached to the baby's wrist.The evaluation will be done while the baby is in the mother's arms, 5 minutes after being placed on the phototherapy bed, and at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st and 24th hours after being placed on the phototherapy bed.
Stress level | mother's arms, 5 minutes after the baby is placed in the phototherapy bed, 5 minutes after the baby is placed in the phototherapy bed at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, and 24th hours.
  Stress level in babies is evaluated with the "Newborn Stress Scale", whose Cronbach's alpha coefficient is between 0.65-0.81. The scale is a 3-point Likert type with a total of 24 items consisting of 8 sub-dimensions: facial expression, body color, respiration, activity level, consolability, muscle tone, extremities and posture. The items in the scale are graded according to the stress level and classified into 8 subgroups. Each subgroup is evaluated between 0-2 points, and a minimum of 0 and a maximum of 16 points are obtained from the scale. A score of 0 from the baby indicates that the baby's condition is stable and balanced. A high total score on the scale indicates that the baby's stress level is high. The evaluation will be done while the baby is in the mother's arms, 5 minutes after being placed on the phototherapy bed, and at the 3rd, 6th, 9th, 12th, 15th, 18th, 21st and 24th hours after being placed on the phototherapy bed.
Blood bilirubin level | 18th and 24th hours
  The blood bilirubin level of all babies observed for 24 hours, measured in line with the clinical routine, was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ahu Pınar TURAN, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I Don't Plan to Share IPD

REFERENCES:
- [Background] Chen J, Sadakata M, Ishida M, Sekizuka N, Sayama M. Baby massage ameliorates neonatal jaundice in full-term newborn infants. Tohoku J Exp Med. 2011 Feb;223(2):97-102. doi: 10.1620/tjem.223.97. PMID 21263210
- [Background] Chey WY, Lee KY. Motilin. Clin Gastroenterol. 1980 Sep;9(3):645-56. No abstract available. PMID 7000397
- [Background] Ceylan SS, Bolısık B. Examining the psychometric properties of the neonatal stress scale. Acıbadem University Journal of Health Sciences. 2017; (2):97-103.
- [Background] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Background] Dur S, Gozen D. Nonnutritive Sucking Before Oral Feeding of Preterm Infants in Turkey: A Randomized Controlled Study. J Pediatr Nurs. 2021 May-Jun;58:e37-e43. doi: 10.1016/j.pedn.2020.12.008. Epub 2021 Jan 6. PMID 33422394
- [Background] Gozen D, Yilmaz OE, Dur S, Caglayan S, Tastekin A. Transcutaneous bilirubin levels of newborn infants performed abdominal massage: A randomized controlled trial. J Spec Pediatr Nurs. 2019 Apr;24(2):e12237. doi: 10.1111/jspn.12237. Epub 2019 Feb 28. PMID 30817090
- [Background] Hamosh M. A review. Fat digestion in the newborn: role of lingual lipase and preduodenal digestion. Pediatr Res. 1979 May;13(5 Pt 1):615-22. doi: 10.1203/00006450-197905000-00008. No abstract available. PMID 382069
- [Background] Kundt G. A new proposal for setting parameter values in restricted randomization methods. Methods Inf Med. 2007;46(4):440-9. doi: 10.1160/me0398. PMID 17694238
- [Background] Lubbe W, Ten Ham-Baloyi W. When is the use of pacifiers justifiable in the baby-friendly hospital initiative context? A clinician's guide. BMC Pregnancy Childbirth. 2017 Apr 27;17(1):130. doi: 10.1186/s12884-017-1306-8. PMID 28449646
- [Background] Mitra S, Rennie J. Neonatal jaundice: aetiology, diagnosis and treatment. Br J Hosp Med (Lond). 2017 Dec 2;78(12):699-704. doi: 10.12968/hmed.2017.78.12.699. PMID 29240507
- [Background] Nyqvist KH, Haggkvist AP, Hansen MN, Kylberg E, Frandsen AL, Maastrup R, Ezeonodo A, Hannula L, Haiek LN; Baby-Friendly Hospital Initiative Expert Group. Expansion of the baby-friendly hospital initiative ten steps to successful breastfeeding into neonatal intensive care: expert group recommendations. J Hum Lact. 2013 Aug;29(3):300-9. doi: 10.1177/0890334413489775. Epub 2013 May 31. PMID 23727630
- [Background] Montealegre A, Charpak N, Parra A, Devia C, Coca I, Bertolotto AM. [Effectiveness and safety of two phototherapy devices for the humanised management of neonatal jaundice]. An Pediatr (Engl Ed). 2020 Feb;92(2):79-87. doi: 10.1016/j.anpedi.2019.02.008. Epub 2019 Apr 9. Spanish. PMID 30979682
- [Background] Widstrom AM, Marchini G, Matthiesen AS, Werner S, Winberg J, Uvnas-Moberg K. Nonnutritive sucking in tube-fed preterm infants: effects on gastric motility and gastric contents of somatostatin. J Pediatr Gastroenterol Nutr. 1988 Jul-Aug;7(4):517-23. doi: 10.1097/00005176-198807000-00007. PMID 2899621
- [Background] World Health Organizations. Protecting, Promoting And Supporting Breastfeeding In Facilities Providing Maternity And Newborn Services: The Revised Baby-Friendly Hospital Initiative, 2018. https://apps.who.int/iris/bitstream/handle/10665/272943/9789241513807-eng.pdf, [Access Address: 21 February 2024].